CLINICAL TRIAL: NCT03551925
Title: Effect of Occupational Therapy in Promoting Medication Adherence: A Randomized Control Trial
Brief Title: Effect of Occupational Therapy in Promoting Medication Adherence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Indianapolis (Other)
Collaborators: University of Missouri, Kansas City (Other); Missouri State University (Other)
Responsible Party: Principal Investigator, Elizabeth Moore, Assistant Professor, Co-Chair Human Research Protections Program, University of Indianapolis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0901
Record Dates: First submitted 2018-05-26; First posted 2018-06-11 (Actual); Last update posted 2019-06-18 (Actual); Status verified 2019-06

CONDITIONS: Hypertension; Diabete Type 2
MeSH Terms: conditions — Hypertension; Diabetes Mellitus, Type 2 | interventions — Therapeutics; Occupational Therapy

STUDY DESIGN:
Intervention Model Description: This will be a randomized controlled trial using a pretest-posttest control group design to allow for comparison between a treatment as usual (TAU) group supporting medication adherence and a TAU group that receives an additional occupational therapy intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment as Usual Plus Occupational Therapy (Experimental): The occupational therapy intervention will be guided by the Integrative Medication Self-Management Intervention (IMedS).The IMedS process guides the occupational therapist and client through an initial evaluation process and a three-step intervention plan to improve medication management.
  Interventions: Behavioral: Treatment as Usual Plus Occupational Therapy
- Treatment as Usual (TAU) (Active Comparator): Participants will receive only the TAU intervention which is provided by a clinical pharmacist and is the protocol at Jordan Valley Community Health Center. The intervention seeks to improve medication adherence in individuals with hypertension.
  Interventions: Behavioral: Treatment as Usual

INTERVENTIONS:
Behavioral: Treatment as Usual Plus Occupational Therapy — The IMeds consists of a three-step process that leads the client from the reflection of past performance, to goal setting, and onto strategy identification and implementation. This intervention guides the client through identifying strategies in the following six areas: altering the medication management activity, advocacy, assistive technology, environmental modifications, and securing refills on time (Schwartz et al., 2017).
  Other Names: IMeds
  Arms: Treatment as Usual Plus Occupational Therapy
Behavioral: Treatment as Usual — A clinical pharmacist counsels participants on proper medication adherence.
  Arms: Treatment as Usual (TAU)

SUMMARY:
The purpose of this research study is to see if an occupational therapist can help people with high blood pressure and/or diabetes find ways to better take their medicine. Participants will be recruited from the Jordan Valley Community Health Center in Springfield, Missouri.

DETAILED DESCRIPTION:
The purpose of this study is to determine whether the addition of an occupational therapy intervention to counseling by a clinical pharmacist (current usual care) compared to counseling by a clinical pharmacist only, will affect three-month medication adherence rates among community-dwelling adults with uncontrolled hypertension and/or diabetes.

To meet this purpose, the following objectives will be addressed:

1. to determine if the addition of the delivery of an occupational therapy intervention (specifically the Integrative Self-Management Intervention) to usual care improves three-month medication adherence rates, as measured by the Adherence to Refills and Medication Scale (ARMS-7), pill count, blood pressure and/or hemoglobin A1c.
2. to determine whether the administration of the occupational therapy intervention in addition to usual care influences an individual's readiness for change as measured by the stages of change measure; and
3. to explore whether participant demographics (e.g., gender, age, race/ethnicity, assist at home, co-morbidities, and number of medications) impact three-month medication adherence rates.

ELIGIBILITY:
Inclusion Criteria:

* Jordan Valley Community Health Center clients will be considered eligible for inclusion in the study if they are 18 years or older, have a confirmed diagnosis of hypertension, receive a score of less than or equal to 21 on the Adherence to Refills and Medication Scale (ARMS-7) and they provide written informed consent.

Exclusion Criteria:

* Participants will be excluded if they indicate via self-report that they are unable to read or understand spoken English without an interpreter or translator or if they have a medical power of attorney and are unable to provide their own informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
Change in Adherence to Refills and Medication Scale (Seven-item) (ARMS-7) Score | The ARMS-7 will be given approximately every 4 weeks over a 12 week period by the clinical pharmacist.
  The ARMS-7 consists of seven questions that provide a self-report of medication adherence.

SECONDARY OUTCOMES:
Change in Stages of Change Measure Score | The stages of change measure will be given approximately every 4 weeks over a 12 week period by the clinical pharmacist.
  A single-item multiple choice question that assesses an individuals current readiness for change.
Change in Pill count | Pill count will be completed approximately every 4 weeks over a 12 week period by the clinical pharmacist.
  A percentage of adherence can be calculated by pill count which includes dividing the number of doses taken by the number of doses that should have been taken multiplied by 100.
Change in Blood pressure | Blood pressure will be taken approximately every 4 weeks over a 12 week period by the clinical pharmacist.
  Use of the manual auscultatory method for taking blood pressure will be completed by the clinical pharmacist. Systolic and diastolic blood pressures will be recorded and compared separately.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Moore, PhD, Principal Investigator — University of Indianapolis
Locations (1):
- Jordan Valley Community Health Center, Springfield, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schwartz JK, Grogan KA, Mutch MJ, Nowicki EB, Seidel EA, Woelfel SA, Smith RO. Intervention to Improve Medication Management: Qualitative Outcomes From a Phase I Randomized Controlled Trial. Am J Occup Ther. 2017 Nov/Dec;71(6):7106240010p1-7106240010p10. doi: 10.5014/ajot.2017.021691. PMID 29135431